CLINICAL TRIAL: NCT01431807
Title: An Open-label, Multicenter, Long-term Phase 3 Study to Evaluate the Safety and Efficacy of Long-term Treatment With SYR-472 in the Treatment of Type 2 Diabetes Mellitus With Inadequate Glycemic Control Despite Diet and/or Exercise Therapies or Treatment With an Existing Oral Anti-diabetic Drug Added to Diet and/or Exercise Therapies
Brief Title: Long-term Study of SYR-472
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYR-472/OCT-001; JapicCTI-111592 (Registry Identifier: JapicCTI); U1111-1123-6415 (Registry Identifier: WHO)
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — trelagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYR-472 group (Experimental): (long-term monotherapy or long-term combination therapy with anti-diabetic drugs)
  Interventions: Drug: SYR-472

INTERVENTIONS:
Drug: SYR-472 — oral, for up to 52 weeks.

SUMMARY:
To evaluate the safety and efficacy of long-term treatment with SYR-472 in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is an outpatient.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Diabetes Mellitus

Exclusion Criteria:

1. The participant has any serious cardiac disease, serious cerebrovascular disorder, or any serious pancreatic or hematological disease.
2. The participant is considered ineligible for the study for any other reason by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Takeda (Note: This product was divested to Teijin Pharma Limited in 2023)
Locations (41):
- Japan (41):
  - Akita, Akita
  - Kisarazu-shi, Chiba
  - Fukuoka, Fukuoka
  - Munakata-shi, Fukuoka
  - Koriyama-shi, Fukushima
  - Gihu-shi, Gihu
  - Fukuyama-shi, Hiroshima
  - Hiroshima, Hiroshima
  - Eniwa-shi, Hokkaido
  - Ishikari-shi, Hokkaido
  - Nakagawa-gun, Hokkaido
  - Obihiro-shi, Hokkaido
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Mito, Ibaragi
  - Naka, Ibaragi
  - Takamatsu, Kagawa-ken
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Tamana-shi, Kumamoto
  - Kyoto, Kyoto
  - Nagano, Nagano
  - Nagawaki-shi, Nagasaki
  - Ōita, Oita Prefecture
  - Minoh, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Ageo-shi, Saitama
  - Kawaguchi-shi, Saitama
  - Koshigaya-shi, Saitama
  - Kuki-shi, Saitama
  - Saitama-shi, Saitama
  - Suntou-gun, Shizuoka
  - Oyama-shi, Tochigi
  - Chuo-ku, Tokyo
  - Koganei-shi, Tokyo
  - Meguro-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Tama-shi, Tokyo
  - Tiyoda-ku, Tokyo